CLINICAL TRIAL: NCT04874454
Title: Evaluating Potential Risk of Choking by Laryngeal Ultrasound in Patients With Acute Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 202101143RINA
Record Dates: First submitted 2021-05-02; First posted 2021-05-05 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Acute Stroke
MeSH Terms: conditions — Stroke | interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- vocal cord movement among the stroke patients (Experimental)
  Interventions: Diagnostic Test: ultrasound

INTERVENTIONS:
Diagnostic Test: ultrasound — evaluate the vocal cord movement among the stroke patients

SUMMARY:
The investigators evaluate the vocal cord movement in patients with acute stroke by ultrasound. The occurrence of choking or aspiration pneumonia will be collected in one year after the index stroke.

DETAILED DESCRIPTION:
Post-stroke dysphagia is a common complication for the stroke patient. It may cause aspiration, poor nutrition or even pneumonia; thus, it is crucial for the physicians to evaluate the swallowing function of the stroke patients. However, the evaluation methods nowadays still have some limitations. Water swallowing test is one of the well-known methods, but the test itself would put the patients at risk of aspiration. Furthermore, in order to increase the sensitivity of the water swallowing test, the amount of the water should also be increased; as a consequence, the risk of aspiration will also increase. Fiberoptic endoscopic evaluation of the swallowing and videofluoroscopy have limitations of invasiveness. The laryngeal ultrasound to evaluate the vocal cord movement can be an alternative method, having the characteristics of non-invasiveness and repeat evaluation.

The investigators aim to evaluate the vocal cord movement in patients with acute stroke by ultrasound. The occurrence of choking or aspiration pneumonia will be collected in one year after the index stroke.

ELIGIBILITY:
Inclusion Criteria:

* acute stroke (in one month) patients

Exclusion Criteria:

* patients with stroke occurring more than one month ago

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-07-14 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
the incidence of aspiration pneumonia | one year

CONTACTS AND LOCATIONS:
Overall Officials: Wan-Ching Lien, Principal Investigator — National Taiwan University Hospital
Locations (1):
- Wan-Ching Lien, Taipei, None Selected, Taiwan

IPD SHARING:
Plan to Share IPD: No